CLINICAL TRIAL: NCT05776043
Title: Empagliflozin and Dapagliflozin in Patients Hospitalized for Acute Decompensated Heart Failure (EMPATHY) - a Phase III Trial.
Brief Title: Empagliflozin and Dapagliflozin in Patients Hospitalized for Acute Decompensated Heart Failure
Acronym: EMPATHY
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Warsaw (Other)
Collaborators: Medical University of Vienna (Other); Medical University of Graz (Other); University Clinical Center of the Medical University of Warsaw (Unknown); Jerzy Popiełuszko Bielański Hospital in Warsaw (Unknown); Regional Polyclinical Hospital in Kielce (Unknown); University Clinical Hospital Military Medical Academy, Central Veterans Hospital in Łódź (Unknown); Medical University of Gdansk (Other); Autonomous Public Specialist Western John Paul II Hospital in Grodzisk Mazowiecki (Unknown); Nicolaus Copernicus University in Toruń, Collegium Medicum in Bydgoszcz (Other); Poznan University of Medical Sciences (Other); John Paul II Hospital, Krakow (Other); Ludwik Rydygier Regional Polyclinical Hospital in Toruń (Unknown); University Teaching Hospital in Białystok (Unknown); Medical University of Silesia in Katowice (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EMPATHY; 2020-003497-48 (EudraCT Number); 2019/ABM/01/00037 (Other Grant/Funding Number: Medical Research Agency (ABM))
Record Dates: First submitted 2022-04-04; First posted 2023-03-20 (Actual); Last update posted 2023-03-20 (Actual); Status verified 2023-03

CONDITIONS: Acute Decompensated Heart Failure
Keywords: SGLT-2 inhibitors; dapagliflozin; empagliflozin; acute heart failure; decompensated heart failure
MeSH Terms: interventions — empagliflozin; dapagliflozin

STUDY DESIGN:
Intervention Model Description: Two arms with a subsequent stratification based on the SGLT2 inhibitor type.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: double blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- SGLT 2 Inhibitor (Active Comparator): Empagliflozin (n=341) or Dapagliflozin (n=341): 9 months of treatment
  Interventions: Drug: Empagliflozin 10 MG; Drug: Dapagliflozin 10 MG
- Placebo with a switch to SGLT 2 Inhibitor (Placebo Comparator): Placebo (n=682) for 3 months of treatment with a subsequent switch to Empagliflozin (n=341) or Dapagliflozin (n=341): 6 months of treatment
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Empagliflozin 10 MG — once daily for 6 or 9 months
  Other Names: Jardiance
  Arms: SGLT 2 Inhibitor
Drug: Dapagliflozin 10 MG — once daily for 6 or 9 months
  Other Names: Forxiga
  Arms: SGLT 2 Inhibitor
Drug: Placebo — once daily for 3 months
  Other Names: Placebo with switch to SGLT2 inhibitor
  Arms: Placebo with a switch to SGLT 2 Inhibitor

SUMMARY:
National, multicenter, randomized, double-blind, parallel-group, stratified by SGLT-2 inhibitor type, placebo-controlled trial, - a Phase III study. Primary objective of the study is to investigate the impact of SGLT-2 inhibitors (Empagliflozin and Dapagliflozin) on clinical endpoints in patients hospitalized with acute/decompensated HF.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years of age with the capacity to provide written informed consent
* Currently hospitalized for a primary diagnosis of acute/decompensated HF (HFrEF, HFmrEF,HFpEF), including symptoms and signs of fluid overload regardless of ejection fraction or diabetes status
* In patients with HFpEF the diagnosis has to be confirmed according to the current HFpEF definition (by non-invasive testing: evidence of structural or functional changes in the heart as evidenced on echocardiography or by invasive testing as LVEDP assessment or right heart catheterisation).
* Randomized no earlier than 24 hours and up to 10 days after initial presentation while still hospitalized
* Stable as defined by: systolic blood pressure (SBP>100 mmHg for the preceding 6 hours)
* No intensification of IV diuretics within the last 6 hours,
* No use of IV vasodilators within the last 6 hours,
* No use of IV inotropes or levosimendan within the last 24 hours prior to randomization
* Elevated NT-proBNP >600 pg/mL during the current hospitalization in patients with HFrEF and >300 pg/mL in patients with HFmrEF or HFpEF (or above 900 pg/ml if atrial fibrillation is present at admission independently from EF).
* eGFR >20 ml/min/1,73m2

Exclusion Criteria:

* History of ketoacidosis
* Type 1 diabetes
* SGLT-2 Inhibitor at baseline or known allergy to SGLT-2 Inhibitors
* Current active cancer with less than 2 years of life expectancy
* Pulmonary embolism, cerebrovascular accident as the primary trigger for the current hospitalization
* Cardiomyopathy based on infiltrative diseases (e.g. amyloidosis), accumulation diseases (e.g. haemochromatosis, Fabry disease), muscular dystrophies, cardiomyopathy with reversible causes (e.g. stress cardiomyopathy), hypertrophic obstructive cardiomyopathy or known pericardial constriction
* Any severe (obstructive or regurgitant) valvular heart disease, expected to lead to surgery during the trial period
* Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant
* Blood pH<7.32
* >1 episode of severe hypoglycaemia within the last 6 months under treatment with insulin or sulfonylurea
* Acute symptomatic urinary tract infection or genital infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1364 (Estimated)
Dates: Start 2022-03-15 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Time to first event of adjudicated cardiovascular (CV) death, or adjudicated hospitalization for heart failure in patients with heart failure with reduced ejection fraction (HFrEF) | at 3 and 9 months
  combined endpoint

SECONDARY OUTCOMES:
Difference in the number of recurrent hospitalizations due to heart failure between the treatment groups | at 3 and 9 months
  recurrent hospitalizations due to heart failure
Difference in the number of hospitalizations for CV causes between the treatment groups | at 3 and 9 months
  hospitalizations for CV causes
Difference in the number of hospitalizations for other than CV causes between the treatment groups | at 3 and 9 months
  hospitalizations for other than CV causes
Time to adjudicated CV death | at 3 and 9 months
  CV death
Time to adjudicated all cause death | at 3 and 9 months
  all cause death
Time to adjudicated myocardial infarction | at 3 and 9 months
  myocardial infarction
eGFR (Estimated Glomerular Filtration Rate) (CKD-EPI (Chronic Kidney Disease Epidemiology Collaboration Equation)) creatine slope of change from baseline between the treatment groups | at 3 and 9 months
  eGFR
Difference in the number of hospital re-admissions due to heart failure between the treatment groups | at 3 and 9 months
  hospital re-admissions due to heart failure
Difference in the number of hospital re-admissions for any cause between the treatment groups | at 3 and 9 months
  hospital re-admissions for any cause
Difference in the duration of hospital stay between the treatment groups after initiation of the study treatment | at 3 and 9 months
  duration of hospital stay
Difference in the number of incidences of new onset AF and re-occurrence of AF between treatment groups | at 3 and 9 months
  new onset AF
Difference in the change of ejection fraction in echocardiography between treatment groups | at 3 and 9 months
  ejection fraction
Difference in the change of left ventricular diastolic function in echocardiography | at 3 and 9 months
  left ventricular diastolic function
Difference in the change of LV strain analysis in echocardiography | at 3 and 9 months
  LV strain
The time-averaged proportional change in NT-proBNP from | at 3 and 9 months
  NT-proBNP
The time-averaged proportional change in selected miRNA expression linked to hypertrophy, inflammation, fibrosis, apoptosis, electric stability between treatment groups and placebo group | at 3 and 9 months
  miRNA expression
The time-averaged proportional change in pre-specified biomarkers | at 3 and 9 months
  biomarkers
Change from baseline in clinical summary score (HF (Chronic Heart Failure) symptoms and physical limitations domains) of the Kansas City Cardiomyopathy Questionnaire (KCCQ) | at 3 and 9 months
  HF score

CONTACTS AND LOCATIONS:
Locations (1):
- Autonomous Public Specialist Western John Paul II Hospital, Grodzisk Mazowiecki, Poland